CLINICAL TRIAL: NCT03886662
Title: A Phase 1b/2 Study Evaluating the Safety and Efficacy of Intravenous LB-100 in Patients With Low or Intermediate-1 Risk Myelodysplastic Syndromes (MDS) Who Had Disease Progression or Are Intolerant to Prior Therapy
Brief Title: A Study of LB-100 in Patients With Low or Intermediate-1 Risk Myelodysplastic Syndromes (MDS)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lixte Biotechnology Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19635
Record Dates: First submitted 2019-03-18; First posted 2019-03-22 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — LB100

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LB-100 for Intravenous administration (Experimental): Phase Ib: Escalating doses of LB-100 administered. Phase 2: Safe dose of LB-100 from phase Ib administered.
  Interventions: Drug: LB-100

INTERVENTIONS:
Drug: LB-100 — Phase Ib: Two escalating doses of LB-100 in two separate cohorts will be administered intravenously on days 1, 3 and 5 of a 21-day cycle over 120 minutes.
  Phase 2: Safe dose of LB-100 as determined from phase Ib will be administered intravenously on days 1, 3 and 5 of a 21-day cycle over 120 minutes.

SUMMARY:
The purpose of this study is to test the safety and efficacy (benefits) of an investigational drug LB-100, for treatment of myelodysplastic syndromes. LB-100 has previously been administered to patients with various solid tumors. In this study, LB-100 will be administered as an intravenous infusion over 120 minutes. This study will be conducted in 2 phases. In phase Ib, escalating doses of LB-100 will be administered to patients to study the safety and to determine a safe dose of LB-100. In phase 2, patients will be administered LB-100 at the dose that was found to be safe in phase Ib. The efficacy (benefits) and safety of LB-100 will be determined in this phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the Informed Consent Form (ICF) and is able to comply with protocol requirements.
2. Patient has adequate organ function as defined by the following laboratory values:

   * Creatinine clearance (CrCl) ≥ 60ml/min
   * Total serum bilirubin < 1.5 x Upper Limit of Normal (ULN) or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range only in patients with well documented Gilbert's syndrome or hemolysis or who required regular blood transfusions
   * Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) < 3.0 x ULN
3. Age ≥18 years at the time of signing the informed consent form.
4. Documented diagnosis of MDS or MDS/myeloproliferative neoplasm (MPN) by World Health Organization (WHO) criteria that require treatment due to cytopenias and meet the International Prognostic Scoring System (IPSS) criteria for low or int-1 risk.
5. For non-del(5q) patients, failed prior treatment with at least 2 cycles started of azacitidine or decitabine or lenalidomide defined as no response to treatment, loss of response at any time point while on treatment or within 6 months of treatment discontinuation, or progressive disease/intolerance to therapy.
6. For del(5q) patients, failed prior treatment with at least 2 cycles started of lenalidomide defined as no response to treatment, loss of response at any time point, or progressive disease/intolerance to therapy.
7. An Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
8. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence; tubal ligation, partner's vasectomy) prior to Cycle 1 Day 1 (C1D1) and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

1. Patient has a known history of HIV infection (testing not mandatory).
2. Patient has any of the following cardiac abnormalities:

   * symptomatic congestive heart failure
   * myocardial infarction ≤ 6 months prior to enrollment
   * unstable angina pectoris as designated by the treating physician
   * serious uncontrolled cardiac arrhythmia as designated by the treating physician
   * QTcF (Fridericia's correction formula) ≥ 450 msec
3. Concomitant malignancies or previous malignancies with less than a 1-year disease free interval at the time of enrollment. Patients with adequately resected basal or squamous cell carcinoma of the skin, or adequately resected carcinoma in situ (i.e. cervix) may enroll irrespective of the time of diagnosis.
4. Use of chemotherapeutic agents or experimental agents (agents that are not commercially available) for the treatment of MDS within 14 days of the first day of study drug treatment.
5. No concurrent use of erythroid stimulating agents, Granulocyte-colony stimulating factor (G-CSF), Granulocyte-macrophage colony-stimulating factor (GM-CSF) is allowed during study except in cases of febrile neutropenia where G-CSF can be used for short term. Growth factors must be stopped two weeks prior to study.
6. Pregnant women are excluded from this study because LB-100 has not been studied in pregnant subjects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LB-100, breastfeeding should be discontinued if the mother is treated with LB-100.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
For Phase Ib - Number of patients with adverse events related to the study treatment as a measure of safety and tolerability of LB-100 study drug | From the first dose of the study drug to 30-days following last dose of the study drug
  Number of patients with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events v5.0 (CTCAE v5.0)
For Phase 2 - Best overall response rate of patients to the study treatment as a measure of efficacy of LB-100 study drug | At screening and then at the end of Cycle 3 and Cycle 6. (Each cycle is 21 days)
  Best overall response rate of the patients to the study treatment as assessed by International Working Group (IWG) 2006 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Rami Komrokji, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States